CLINICAL TRIAL: NCT01813344
Title: The Clinical Outcomes of Hyper-CVAD Treatment in Lymphoblastic Lymphoma
Brief Title: Hyper-CVAD Treatment in Lymphoblastic Lymphoma
Acronym: LBL-CISL-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Seong Hyun Jeong, Assistant professor, Ajou University School of Medicine
Other Study IDs: LBL-CISL-1
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Lymphoblastic Lymphoma
Keywords: Adult lymphoblastic lymphoma; Hyper-CVAD; first-line treatment
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Treatment outcomes of lymphoblastic lymphoma (LBL) have improved by the use of the regimens for acute lymphoblastic leukemia. Hyper-CVAD is one of the most effective treatments with high remission rate in acute lymphoblastic leukemia (ALL) and LBL. However, the treatment outcome of hyper-CVAD in LBL has reported only in small number of patients from single institution. The investigators conducted this study to evaluate the hyper-CVAD regimen based treatment in LBL.

DETAILED DESCRIPTION:
We will analyze treatment outcome of lymphoblastic lymphoma patients treated with hyper-CVAD regimen from 13 institutions in Korea. In all patients, hyper-CVAD was initial treatment. After achievement of response, patients either underwent hematopoietic stem cell transplantation (HSCT) or consolidation with hyper-CVAD.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 at diagnosis
* Pathologically proven lymphoblastic lymphoma

Exclusion Criteria:

* proven HIV infection
* pretreatment with other regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult lymphoblast lymphoma patients treated with hyper-CVAD regimen in Korea
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3-year
Progression free survival | 3-year

SECONDARY OUTCOMES:
Response Rate | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou Universtiy School of Medicine, Suwon, Kyeonggi, South Korea